CLINICAL TRIAL: NCT03194594
Title: The Effects of Combination of Intravenous Dexamethasone and Ketamine on Change of Postoperative Mood in Patients Undergoing Laparoscopically Assisted Gynecologic Surgery.
Brief Title: Dexamethasone and Ketamine on Change of Postoperative Mood
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Cheol Lee, Chief professor, principal investigator, Wonkwang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WonkwangUH2
Record Dates: First submitted 2017-06-13; First posted 2017-06-21 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Depressive Symptoms
Keywords: Ketamine, dexamethasone, mood
MeSH Terms: conditions — Depression | interventions — Ketamine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group K (n = 31) (Active Comparator): will receive a single dose of ketamine 0.5 mg/kg i.v. plus 2 ml normal saline, at 5 minutes after the induction of anesthesia
  Interventions: Drug: Ketamine Hydrochloride, dexamethasone, and combination of two drugs
- Group D (n = 31) (Active Comparator): will receive dexamethasone 0.5 mg/kg i.v. plus 2 ml normal saline, at 5 minutes after the induction of anesthesia
  Interventions: Drug: Ketamine Hydrochloride, dexamethasone, and combination of two drugs
- Group KD (n = 31) (Experimental): will receive ketamine 0.5 mg/kg i.v. and dexamethasone 0.5 mg/kg i.v., at 5 minutes after the induction of anesthesia
  Interventions: Drug: Ketamine Hydrochloride, dexamethasone, and combination of two drugs

INTERVENTIONS:
Drug: Ketamine Hydrochloride, dexamethasone, and combination of two drugs — After receiving by IRB approval and obtaining informed consent from patients, 93 patients who were aged between 18 and 70 years old and classified as American Society of Anesthesiologists (ASA) classes I and II. Afterward, the patients are randomly (sealed envelopes) allocated into one of three treatment; Group K (n = 31) receives a single dose of ketamine 0.5 mg/kg i.v. plus 2 ml normal saline, Group D (n = 31) receives dexamethasone 0.5 mg/kg i.v. and a maximum dose of 8 mg plus 2 ml saline, and Group KD (n = 31) receiveds ketamine 0.5 mg/kg i.v. and dexamethasone 0.5 mg/kg i.v. at 5 minutes after the induction of anesthesia in a double-blinded method.

SUMMARY:
Ketamine and dexamethasone have been known to be effective postoperative pain. Many studies also have reported these two drugs might change mood such as depression. This study aimed to investigate the effect of each drug individually with their combination on perioperative change of mood in patients undergoing gynecologic surgery

DETAILED DESCRIPTION:
After receiving by IRB approval and obtaining informed consent from patients, 93 patients who are aged between 18 and 70 years old and classified as American Society of Anesthesiologists (ASA) classes I and II.

Afterward, the patients will be randomly (sealed envelopes) allocated into one of three treatment; Group K (n = 31) will receive a single dose of ketamine 0.5 mg/kg i.v. plus 2 ml normal saline, Group D (n = 31) receive dexamethasone 0.5 mg/kg i.v. and a maximum dose of 8 mg plus 2 ml saline, and Group KD (n = 31) receive ketamine 0.5 mg/kg i.v. and dexamethasone 0.5 mg/kg i.v. at 5 minutes after the induction of anesthesia in a double-blinded method.

ELIGIBILITY:
A total of 93 patients

Inclusion Criteria:

* patients who were scheduled for laparoscopic gynecologic surgery

Exclusion Criteria:

* Patients with hepatic and renal insufficiency, history of allergy to the study drugs, previous gastric ulcer, diabetes mellitus, and receiving analgesic, antiemetic, antihistamine, steroids or psychiatric drugs within 24 hours before surgery steroids

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-12 (Actual)

PRIMARY OUTCOMES:
The change of patient health questionnaire (PHQ)-9 scores | at the 1st day after surgery
  Anesthesiologist performed the assessment of perioperative depressed mood change with use of Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is the depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day) with a total score ranging from 0 to 27; 0-4 none, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe depressed mood

SECONDARY OUTCOMES:
postoperative visual analog scale (VAS) for pain | for 48 h after surgery
  The VAS consisted of a straight line with the left end of the line representing no pain and the right end of the line representing the worst pain. Patients were asked to mark the position on the line corresponding to their perception of pain. The VAS score for pain was measured with intervals of 1, 6, 24, and 48 hours after surgery.
patient controlled analgesia (PCA) consumption | for 24 h after surgery
  Each patient was administered analgesics using a PCA pump containing morphine (60 mg), ketorolac (150 mg), and ramosetron (0.6 mg) in a total volume of 100 ml of saline. This device was set to deliver a basal infusion of 2 ml/hr and bolus doses of 0.5 ml with a 15 min lockout period.

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Lee, M.D.,Ph.D, Principal Investigator — Wonkwang UH
Locations (1):
- WonwangUH, Iksan, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided